CLINICAL TRIAL: NCT03885037
Title: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" General Investigation (Rheumatoid Arthritis)
Brief Title: Infliximab Biosimilar for Intravenous Drip Infusion 100 mg "Pfizer" Drug Use Investigation (Rheumatoid Arthritis)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B5371006; NCT03885037 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-03-04; First posted 2019-03-21 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Infliximab; biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab [infliximab biosimilar 3]: Patients with Rheumatoid Arthritis treated by Infliximab BS
  Interventions: Drug: Infliximab [infliximab biosimilar 3]

INTERVENTIONS:
Drug: Infliximab [infliximab biosimilar 3] — <Rheumatoid arthritis> The usual dose is 3 mg as Infliximab [Infliximab Biosimilar 3] for every kg of body weight given as an intravenous infusion. After an initial dose is given, the subsequent doses are given at Weeks 2 and 6, and every 8 weeks thereafter. After a dose at Week 6 is given, the dose may be increased or the dosing interval may be reduced for patients who have an incomplete response or reduced effects. These adjustments should be made in a stepwise manner. The maximum dose is 10 mg for every kg of body weight at the dosing interval of 8 weeks and 6 mg for every kg of body weight at a reduced dosing interval. The minimum dosing interval is 4 weeks. This drug should be given in combination with methotrexate.
  Other Names: Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer"

SUMMARY:
To collect information on the safety and effectiveness of Infliximab BS for Intravenous Drip Infusion 100 mg "Pfizer" against rheumatoid arthritis under actual status of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis who started treatment with this drug
* Patients who received this drug for the first time after the day of launch of this drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis treated by Infliximab BS
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5371006

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]: Participants with rheumatoid arthritis (RA) who received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] as indicated in the approved local product document for the first time were observed for 30 weeks from the day of initial dose of this drug. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Started | 77
Completed | 61
Not Completed | 16
Not completed — Protocol Violation | 16

BASELINE CHARACTERISTICS:
Population: A total of 77 participants were enrolled in this study. Of the 77 participants from whom case report forms were collected, 16 participants were excluded due to protocol violation. The remaining 61 participants were included in the safety analysis set.
Groups:
- Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]: Participants with RA who received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] as indicated in the approved local product document for the first time were observed for 30 weeks from the day of initial dose of this drug. The dosage can be adjusted as per physician's discretion.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 61
Age, Customized [Number; unit: participants]
  <15 years | 0
  ≥15 and <65 years | 29
  ≥65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: An ADR was a treatment-related adverse event, and any untoward medical occurrence attributed to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] in a participant who received this drug. A serious ADR was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; and congenital anomaly/birth defect. Relatedness to Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] was assessed.
Time Frame: 30 weeks from the day of initial dose
Population: The safety analysis set (61 participants) comprised of participants who satisfied the inclusion criteria and had received Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]. Participants with protocol violation were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 61
Participants
  ADR | 3
  serious ADR | 1

2. Secondary Outcome: Change in Disease Activity Score Based on 28-joint Count and C-reactive Protein (4 Variables) (DAS28 [4/CRP])
Description: The Disease Activity Score based on 28-joint count and C-reactive protein (DAS28 [4/CRP]) was calculated using four variables: Tender Joint Count (TJC28) and Swollen Joint Count (SJC28), both scored from 0 to 28; participant's overall activity assessed by the Visual Analog Scale (VAS, 0-100 mm); and C-reactive protein (CRP, ≥0 mg/dL). Higher scores indicate increased disease activity.
  The formula is:
  DAS28 (4/CRP) = 0.56 × √(TJC28) + 0.28 × √(SJC28) + 0.36 × LN((CRP) × 10 + 1) + 0.014 × (VAS) + 0.96.
  Changes in DAS28 (4/CRP) from baseline to study completion were summarized as mean ± standard deviation, overall, as well as separately based on prior infliximab use before the initial dose of this drug. Greater negative changes reflect larger reductions in disease activity.
Time Frame: 30 weeks from the day of initial dose
Population: The efficacy analysis set (54 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 54 participants, 41 participants who had DAS28 (4/CRP) available both at baseline and study completion were evaluated the disease activity at the time of study completion.
  Among the 41 participants, 28 had no prior use of infliximab products, while 13 had used them before.
Measure: Mean (Standard Deviation); unit: Scores of DAS28 (4/CRP)
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 41
Scores of DAS28 (4/CRP)
  Change in DAS28 (4/CRP): overall | -0.864 (1.534)
  Change in DAS28 (4/CRP): no prior infliximab use: number analyzed (Participants) | 28
  Change in DAS28 (4/CRP): no prior infliximab use | -1.184 (1.715)
  Change in DAS28 (4/CRP): prior infliximab use: number analyzed (Participants) | 13
  Change in DAS28 (4/CRP): prior infliximab use | -0.175 (0.689)

3. Secondary Outcome: Percentage of Participants With Remission (DAS28 [4/CRP])
Description: Percentage of participants with a remission based on DAS28 (4/CRP) was presented along with the two-sided 95% confidence interval (exact method).
  For participants with available DAS28 (4/CRP) values both at baseline and study completion, the number and proportion of those who achieved remission (<2.3) at both time points were calculated overall, as well as separately based on prior infliximab use before the initial dose of this drug.
Time Frame: 30 weeks from the day of initial dose
Population: The efficacy analysis set (54 participants) comprised of participants in the safety analysis set who had effectiveness evaluation. Of the 54 participants, the percentage of participants who achieved remission (< 2.3) as of the study completion date was calculated for the 41 participants whose DAS28 (4/CRP) were available both at baseline and study completion.
  Among the 41 participants, 28 had no prior use of infliximab products, while 13 had used them before.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
Number analyzed (Participants) | 41
Percentage of Participants
  Remission at baseline (overall) | 36.6 [22.12 to 53.06]
  Remission at baseline (no prior infliximab use): number analyzed (Participants) | 28
  Remission at baseline (no prior infliximab use) | 25.0 [10.69 to 44.87]
  Remission at baseline (prior infliximab use): number analyzed (Participants) | 13
  Remission at baseline (prior infliximab use) | 61.5 [31.58 to 86.14]
  Remission at study completion date (overall) | 61.0 [44.50 to 75.80]
  Remission at study completion date (no prior infliximab use): number analyzed (Participants) | 28
  Remission at study completion date (no prior infliximab use) | 53.6 [33.87 to 72.49]
  Remission at study completion date (prior infliximab use): number analyzed (Participants) | 13
  Remission at study completion date (prior infliximab use) | 76.9 [46.19 to 94.96]

ADVERSE EVENTS:
Time Frame: 30 weeks from the day of initial dose
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3]
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 1/61
Other Adverse Events (participants affected / at risk) | 2/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] (N=61)
Altered state of consciousness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab BS for I.V. Infusion 100mg [Pfizer] [Infliximab Biosimilar 3] (N=61)
Herpes zoster (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03885037/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03885037/SAP_001.pdf